CLINICAL TRIAL: NCT07398924
Title: Comparison of Vaginal Estradiol and Oral Guaifenesin Interventions in Patients Undergoing Ovulation Induction With Clomiphene Citrate
Brief Title: Vaginal Estradiol and Oral Guaifenesin in Clomiphene Ovulation Induction
Acronym: CC-OVI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Gamze Karababa, Medical Doctor, Yuzuncu Yil University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: YYU-CC-OVI-2022; YYU-ETH-2021 (Other: Yuzuncu Yil University Ethics Committee Approval)
Record Dates: First submitted 2026-01-26; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Female Infertility; Anovulatory Infertility; Unexplained Infertility
Keywords: Clomiphene citrate, Ovulation induction, Vaginal estradiol, Guaifenesin, Endometrial thickness, Cervical mucus, Infertility treatment
MeSH Terms: conditions — Infertility, Female | interventions — Clomiphene; Guaifenesin; Acetylcysteine; Estradiol; segesterone acetate and ethinyl estradiol vaginal system

STUDY DESIGN:
Intervention Model Description: Participants were randomized into three parallel treatment arms and followed prospectively for outcome assessment.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors were blinded to treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Clomiphene Citrate + Guaifenesin (Experimental): Participants received clomiphene citrate for ovulation induction combined with oral guaifenesin during the follicular phase.
  Interventions: Drug: Clomiphene Citrate.; Drug: Guaifenesin
- Clomiphene Citrate + Vaginal Estradiol (Experimental): Participants received clomiphene citrate for ovulation induction combined with vaginal estradiol during the follicular phase.
  Interventions: Drug: Clomiphene Citrate.; Drug: Estradiol (E2)
- Clomiphene Citrate + Guaifenesin + Vaginal Estradiol (Experimental): Participants received clomiphene citrate combined with both oral guaifenesin and vaginal estradiol during the follicular phase.
  Interventions: Drug: Clomiphene Citrate.; Drug: Guaifenesin; Drug: Estradiol (E2)

INTERVENTIONS:
Drug: Clomiphene Citrate. — Clomiphene citrate administered orally for ovulation induction according to standard clinical protocols.
  Other Names: Clomifene Citrate
Drug: Guaifenesin — Oral guaifenesin administered during the follicular phase to improve cervical mucus characteristics.
  Other Names: Glyceryl guaiacolate
  Arms: Clomiphene Citrate + Guaifenesin; Clomiphene Citrate + Guaifenesin + Vaginal Estradiol
Drug: Estradiol (E2) — Vaginal estradiol administered during the follicular phase to improve endometrial development.
  Other Names: Vaginal Estradiol
  Arms: Clomiphene Citrate + Guaifenesin + Vaginal Estradiol; Clomiphene Citrate + Vaginal Estradiol

SUMMARY:
Clomiphene citrate is commonly used for ovulation induction; however, it may negatively affect endometrial development and cervical mucus quality, which can reduce pregnancy rates. Various adjunctive treatments have been proposed to overcome these antiestrogenic effects.

This randomized clinical trial aimed to compare the effects of vaginal estradiol and oral guaifenesin, alone or in combination, on endometrial thickness, cervical mucus characteristics, and clinical pregnancy rates in women undergoing ovulation induction with clomiphene citrate.

A total of 90 women with infertility undergoing ovulation induction were randomly assigned to one of three treatment groups: clomiphene citrate plus guaifenesin, clomiphene citrate plus vaginal estradiol, or clomiphene citrate combined with both guaife

DETAILED DESCRIPTION:
This study was designed as a single-center, randomized, parallel-group interventional clinical trial conducted at a university-affiliated tertiary care hospital. Women diagnosed with infertility and scheduled for ovulation induction with clomiphene citrate were eligible for inclusion.

Participants were randomly assigned to one of three treatment arms: clomiphene citrate plus oral guaifenesin, clomiphene citrate plus vaginal estradiol, or clomiphene citrate combined with both oral guaifenesin and vaginal estradiol. Clomiphene citrate was administered according to standard ovulation induction protocols. Adjunctive treatments were initiated during the follicular phase.

Baseline demographic and clinical characteristics were recorded. Follicular development and endometrial thickness were assessed by transvaginal ultrasonography. Cervical mucus characteristics, including spinnbarkeit and cervical mucus score, were evaluated during the periovulatory period. Ovulation was triggered when appropriate follicular criteria were met.

The primary outcome of the study was the clinical pregnancy rate. Secondary outcomes included endometrial thickness, cervical mucus quality, ovulation response, cycle cancellation, and miscarriage rate. Statistical analyses were performed to compare outcomes between treatment groups.

''

ELIGIBILITY:
Inclusion Criteria:

* - Women aged 18 to 40 years
* Diagnosis of infertility
* Indication for ovulation induction with clomiphene citrate
* Regular or irregular menstrual cycles suitable for ovulation induction
* At least one patent fallopian tube
* Normal uterine cavity on ultrasonography
* Male partner with normal or mildly abnormal semen parameters
* Willingness to participate and provide informed consent

Exclusion Criteria:

* - Known hypersensitivity to clomiphene citrate, guaifenesin, or estradiol
* Severe male factor infertility
* Presence of uterine anomalies or intrauterine pathology
* Endocrine disorders affecting ovulation (e.g., uncontrolled thyroid disease, hyperprolactinemia)
* Polycystic ovary syndrome requiring alternative stimulation protocols
* History of recurrent pregnancy loss
* Use of hormonal treatment within the last 3 months

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2022-01-06 (Actual); Primary Completion 2023-06-06 (Actual); Study Completion 2023-06-23 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy rate | From ovulation trigger administration to confirmation of clinical pregnancy by transvaginal ultrasonography within the same treatment cycle (approximately 4-6 weeks).
  Clinical pregnancy was defined as the presence of an intrauterine gestational sac detected by transvaginal ultrasonography.

SECONDARY OUTCOMES:
Endometrial thickness | On the day of ovulation trigger administration (cycle day-specific).
  Endometrial thickness was measured by transvaginal ultrasonography.
Cervical mucus score | During the peri-ovulatory period, from the day before ovulation trigger to the day after ovulation trigger (approximately 2-3 days).
  Cervical mucus quality was evaluated using cervical mucus scoring.
Spinnbarkeit | During the peri-ovulatory period, from the day before ovulation trigger to the day after ovulation trigger (approximately 2-3 days).
  Spinnbarkeit was assessed as an indicator of cervical mucus stretchability.
Miscarriage rate | Up to 12 weeks of gestation
  Miscarriage was defined as pregnancy loss before 12 weeks of gestation.
Cycle cancellation rate | By the end of the treatment cycle (one cycle, approximately 28 days).
  Cycle cancellation was recorded when ovulation induction could not be completed.

CONTACTS AND LOCATIONS:
Overall Officials: Gamze K Karababa, Study Director — VAN YUZUNCU YİL UNİVERCITY
Locations (1):
- Van Yuzuncu Yil University Dursun Odabasi Medical Center, Van, Di̇yarbakir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to ethical and privacy considerations.

REFERENCES:
- See also: Related Info — https://clinicaltrials.gov